CLINICAL TRIAL: NCT00580619
Title: Autonomic Nervous System and Chronic Fatigue Syndrome
Acronym: CFS&ANS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 060662; CRC-1636 (Other: Local CRC); CRC-1705 (Other: Local CRC)
Record Dates: First submitted 2007-12-17; First posted 2007-12-27 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Fatigue Syndrome; Orthostatic Intolerance; Postural Tachycardia Syndrome
Keywords: Chronic fatigue syndrome; Postural tachycardia syndrome; Autonomic nervous system
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Orthostatic Intolerance; Postural Orthostatic Tachycardia Syndrome | interventions — Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (markers of sympathetic activity) (Experimental): To evaluate if the various indices of sympathetic activity (Autonomic Function Testing) differ between patients with chronic fatigue syndrome and postural tachycardia syndrome (CFS-P), and CFS without POTS.
  Interventions: Other: Autonomic Function Testing
- 2 (saline) (Experimental): To test the null hypothesis that there is no difference between two saline therapies (pulse saline vs. sham saline) in improving both the fatigue score and postural tachycardia syndrome.Saline infusions
  Interventions: Other: Saline infusions
- 3 (NO inhibition/ autonomic blockade) (Experimental): Response to nitric oxide inhibition in the presence and absence of an intact autonomic nervous system will be evaluated. L-NMMA trimethaphan will be used for NO inhibition and autonomic blockade, respectively.
  Interventions: Drug: L-NMMA trimethaphan
- 4 (methyldopa) (Active Comparator): The effects of chronic autonomic withdrawal on improving symptoms of chronic fatigue and postural tachycardia syndrome will be evaluated
  Interventions: Drug: methyldopa

INTERVENTIONS:
Other: Autonomic Function Testing — The autonomic function tests include asking the subject to breathe deeply for two minutes and breathing as fast and as hard as they can for 30 seconds, maintaining a handgrip for 3 minutes, breathing against pressure for 15 seconds, placing one hand in ice water for 1 minute and an orthostatic test. All these tests are meant to stimulate the autonomic nervous system to produce changes in blood pressure and heart rate of short duration that reflect how well the involuntary nervous system is working. In addition, a 24-hour blood pressure monitoring and exercise test may be also performed in some subjects.
  Arms: 1 (markers of sympathetic activity)
Other: Saline infusions — The effects of continuous IV infusion or pulse IV administration of saline in increasing total blood volume and fatigue score will be evaluated
  Arms: 2 (saline)
Drug: L-NMMA trimethaphan — Trimethaphan IV infusion for approximately 60 minutes at a dose of 4-6 mg/min L-NMMA IV infusion for approximately 45 minutes at 125, 250, and 500 mg/kg/min for 15 minutes each
  Arms: 3 (NO inhibition/ autonomic blockade)
Drug: methyldopa — Aldomet oral twice a day for 12 weeks
  Other Names: Aldomet
  Arms: 4 (methyldopa)

SUMMARY:
The investigators propose to test the hypothesis that the sympathetic nervous system contributes to the cardiovascular and inflammatory abnormalities present in the chronic fatigue syndrome (CFS) and, in particular in the subset of patients characterized by postural tachycardia syndrome (POTS). CFS and POTS are seen mostly in otherwise normal young women, and are the cause of significant disability. A substantial proportion of patients referred for evaluation of POTS met diagnostic criteria for CFS and, conversely, a subset of patients referred for treatment for CFS have POTS. The investigators hypothesize that sympathetic activation underlies the pathophysiology of patients in whom CFS and POTS overlap (CFS-P).

DETAILED DESCRIPTION:
In Specific Aim 1, the investigators will use state-of-the-art measurements of sympathetic activity (autonomic function tests, response to trimethaphan, direct nerve sympathetic traffic recordings with microneurography, plasma norepinephrine, and intraneuronal metabolites), inflammatory mediators (C-reactive protein, inflammatory cytokines), and oxidative stress (isoprostanes) in patients with CFS-P. It is important that appropriate control groups be included, and we will also study patients with CFS without orthostatic tachycardia, patients with POTS without CFS, and normal controls.

The investigators have documented abnormalities in volume regulation in POTS patients. Hypovolemia can contribute to sympathetic activation and, vice versa, sympathetic activation can contribute to hypovolemia. Interrupting this vicious circle with acute saline infusion is the most effective treatment to improve symptoms in POTS patients. Not surprisingly, many POTS patients followed by the investigators, and CFS patients followed by Dr. David Bell, are using saline pulse therapy as a way to alleviate symptoms. However, the efficacy and safety of this approach has not been proven. The investigators propose to validate this treatment in Specific Aim 2.

This group studies show that nitric oxide is arguably the most important metabolic factor involved in cardiovascular regulation. Abnormalities in nitric oxide have been proposed to contribute to CFS and POTS, but proving this has been challenging in part due to its interaction with the sympathetic nervous system. In Specific Aim 3, the investigators propose to investigate the importance of nitric oxide in CFS-P patients using an experimental approach developed in our laboratory to eliminate nitric oxide/autonomic interactions.

Finally, in Specific Aim 4, they propose a proof-of-concept study to test the hypothesis that sympathetic activation contributes to many of the abnormalities found in CFS patients. If our hypothesis is correct, inhibition of sympathetic tone will result in improvement of the abnormalities described in volume, inflammation, and oxidative stress. More importantly, it will result in symptomatic improvement in these patients. The investigators believe, therefore, that the studies proposed in this application will improve the understanding of the pathophysiology of CFS, and provide a rationale approach to the treatment of this disabling condition.

ELIGIBILITY:
Inclusion Criteria:

* Meet CDC diagnostic criteria of CFS (Fukuda et al., 1994)
* Meet diagnostic criteria of POTS (Raj et al., 2005)
* Age between 18-65 years
* Male and female are eligible (although the majority of patients with CFS-P are female)

Exclusion Criteria:

* Presence of medical conditions that can explain postural tachycardia syndrome (e.g., dehydration, medications)
* Presence of medical or psychiatric conditions known to cause fatigue (Fukuda et al., 1994). Inability to give, or withdrawal of, informed consent
* Inability to acquire or maintain adequate long-term intravenous access (peripheral indwelling catheter, PIC)
* Pregnancy
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol
* Patients who are bedridden or chair-ridden

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | Duration of the intervention

SECONDARY OUTCOMES:
Blood Pressure | Duration of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okamoto LE, Raj SR, Peltier A, Gamboa A, Shibao C, Diedrich A, Black BK, Robertson D, Biaggioni I. Neurohumoral and haemodynamic profile in postural tachycardia and chronic fatigue syndromes. Clin Sci (Lond). 2012 Feb;122(4):183-92. doi: 10.1042/CS20110200. PMID 21906029